CLINICAL TRIAL: NCT06488014
Title: Comparison of the Effect of Preoperative and Postoperative Erector Spina Plan Block and Paravertebral Block on Postoperative Pain in Video Assisted Thoracic Surgery (VATS)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Hatice Güneş, Research assistant, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CYGHG1
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Anesthesia; Nerve Block; Pain, Postoperative; Thoracic Surgery, Video Assisted
Keywords: Anesthesia; Nerve Block; Postoperative PAİN; Video Assisted Thoracic Surgery (VATS)
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group E (Active Comparator): Erector spina plan block : Under USG guidance, local anaesthetic will be administered to the fascial plane between the erector spinae muscle and the transverse process.
  Interventions: Procedure: Erector spina plan block (ESP)
- Group P (Active Comparator): Paravertebral block: USG-guided local anaesthetic administration to the side of the vertebral body close to where the spinal nerves exit from the intervertebral foramen.
  Interventions: Procedure: Paravertebral block

INTERVENTIONS:
Procedure: Erector spina plan block (ESP) — In both groups, the relevant methods will be applied at the level of the surgical incision before the surgical incision (pre-emptive) after the patient is asleep and before the patient wakes up at the end of surgery.
  The dose of local anaesthetic to be administered is the same for both groups.
  Drug content to be administered*: total 25 cc volume (13.5 ml 0.5% bupivacaine + 5 ml 2% lidocaine + 1.5 ml morphine (morphine diluted with 0.9% NaCl to 1mg/ml) + 5 ml 0.9% NaCl) (These doses are the routine doses applied in such surgeries in our clinic)
  * Local anaesthetic drug doses in regional anaesthesia: source: Kirk, P. H. I. I. L. I. I. P. P., & Berde, C. B. (2020). Local anaesthetics. Miller's Anaesthesia. 9th ed. Philadelphia: Elsevier Inc, 878-9.
  Arms: Group E
Procedure: Paravertebral block — In both groups, the relevant methods will be applied at the level of the surgical incision before the surgical incision (pre-emptive) after the patient is asleep and before the patient wakes up at the end of surgery.
  The dose of local anaesthetic to be administered is the same for both groups.
  Drug content to be administered*: total 25 cc volume (13.5 ml 0.5% bupivacaine + 5 ml 2% lidocaine + 1.5 ml morphine (morphine diluted with 0.9% NaCl to 1mg/ml) + 5 ml 0.9% NaCl) (These doses are the routine doses applied in such surgeries in our clinic)
  * Local anaesthetic drug doses in regional anaesthesia: source: Kirk, P. H. I. I. L. I. I. P. P., & Berde, C. B. (2020). Local anaesthetics. Miller's Anaesthesia. 9th ed. Philadelphia: Elsevier Inc, 878-9.
  Arms: Group P

SUMMARY:
The aim of this prospective controlled randomised clinical trial was to identify the analgesic method that is more effective than two different regional analgesia techniques routinely used for pain control after video-assisted thoracic surgery (VATS).

The effects of paravertebral block and erector spina plan (ESP) block on acute pain, need for additional analgesics and incidence of chronic pain after video-assisted thoracic surgery (VATS) will be compared before surgical incision (pre-emptive) and at the end of surgery.

It is aimed to show that ESP block, which is a newer method in the literature, provides equivalent / more effective analgesia with paravertebral block.

DETAILED DESCRIPTION:
Pain after thoracic surgery is common and usually severe due to factors such as surgical incisions, damage to the lung tissue and ribs, and irritation of the pleura and intercostal nerves by the chest tube. Thoracotomy is one of the most painful surgical operations and the incidence of chronic pain has been reported to be approximately 65% in most studies. Video-assisted thoracic surgery (VATS) has become more common in recent years. Compared with open thoracotomy, VATS reduces postoperative pain, morbidity and length of hospital stay, which is associated with a smaller extent of tissue trauma. However, VATS still causes moderate to severe acute postoperative pain and chronic pain with an incidence reported in the range of 25-35%.

Accelerated rehabilitation is important in thoracic surgery. Postoperative outcomes are affected by the patient's ability to get out of bed and participate in physical respiratory therapy exercises. Inadequate analgesia is also directly related with postoperative pulmonary functions. Pain may lead to atelectasis, hypoxaemia and pneumonia as a result of ineffective cough and thus inadequate sputum expulsion.

Pain management after VATS is important because it may reduce postoperative complications. Systemic analgesic methods using intravenous (iv) drugs such as lidocaine, nonsteroidal anti-inflammatory drugs, steroids, alpha2-adrenergic agonists or N-methyl-D-aspartate (NMDA) antagonists and thoracic epidural analgesia, The multimodal analgesia approach in which regional analgesia methods such as paravertebral block, erector spina plan (ESP) block, and serratus anterior plan block are combined is an approach with proven efficacy in recent studies and guidelines. Regional analgesia has the potential to reduce postoperative acute pain and chronic pain and to increase early postoperative recovery.

Although thoracic epidural anaesthesia (TEA) is considered the gold standard for the treatment of postoperative pain in thoracic surgery, the presence of possible side effects such as dura perforation, nerve damage, epidural bleeding, risk of hypotension and urinary retention has shown that VATS may require less invasive analgesia. Thoracic paravertebral block (TPVB) provides unilateral thoracic analgesia comparable to TEA. In addition, it is not only less invasive than TEA, but also can maintain haemodynamic stability and carries a lower risk of complications. According to the Enhanced Recovery After Surgery (ERAS) guidelines and the Procedure-specific postoperative pain Management (PROSPECT) group, TPVB is recommended as the primary method of regional analgesia for thoracic surgery.

Paravertebral local anaesthetic may spread to multiple levels into the epidural and intercostal spaces, blocking the spinal nerve and sympathetics, resulting in segmental block and ipsilateral sympathectomy. Major risks or complications of PVB include pneumothorax, hypotension due to bilateral PVBs, dural puncture and possible risks associated with epidural injections, including epidural abscess, epidural haematoma. In recent years, there has been increasing interest in fascial plane blocks, which involve spreading large amounts of local anaesthetics into the fascial planes through which nerves pass or communicate with other areas containing the nerves of interest. The erector spinae plane block is the most widely investigated fascial plane block that is most suitable for thoracic surgery. It is technically easier to perform and theoretically has lower risks of serious adverse events associated with TEA and PVB, including epidural haematoma or abscess or pneumothorax, and is less likely to cause sympathectomy or hypotension. ESPB targets the facial plane between the erector spinae muscles and the posterior border of the transverse processes, blocking the dorsal branches of the spinal nerves and potentially spreading anteriorly into the adjacent paravertebral and epidural spaces, blocking the ventral rami and sympathetic chain.

In VATS patients, ESPB resulted in lower PACU pain scores in the first six hours, lower opioid consumption and shorter PACU length of stay compared with placebo control. There are mixed data on the efficacy of ESPB compared with PVB. Although two equivalence studies failed to demonstrate any clinically significant difference in postoperative pain scores between PVB and ESPB for VATS, two other clinical trials have shown that PVB provides better analgesia in VATS patients.

Preemptive analgesia is a type of antinociceptive treatment. Its emergence is based on the clinical observations of Crile and experimental studies of Woolf. They demonstrated that various antinociceptive techniques applied pre-injury were more effective in reducing central nervous system sensitisation than those applied post-injury. The putative mechanisms of chronic postoperative pain can be explained as sensitisation of peripheral sensory neurons, neuroplasticity in the central nervous system, and neuropathic signalling in the neuro-immune axis. The aim of preemptive analgesia is to prevent central nervous system sensitisation caused by the incision and the inflammatory process caused by the incision with pain relief interventions starting before surgical incision.

In our clinic, the investigators routinely apply both paravertebral block and erector spina block before and/or after the incision as part of a multimodal analgesia approach. Different anaesthetists may have different preferences in the choice of field block. In this study, the investigators planned to investigate the effects of paravertabral block and erector spina plan block before and after VATS on postoperative pain scores and prevention of chronicity of pain.

RESEARCH DESİGN

* Primary Endpoint : Lower pain scores with erector spina plan block in acute post-thoracoscopy pain control
* Secondary Endpoint : Less chronic pain with erector spina plan block

METHOD

VATS (Video Assisted Thoracic Surgery) patients who give consent to the study in the preoperative evaluation and meet the inclusion criteria will be included in the study.

Patients will be grouped according to the analgesia method applied. Demographic data of patients who meet the inclusion criteria will be recorded. Routine ASA monitoring: ECG, fingertip saturation, noninvasive blood pressure, neuromuscular junction monitoring (TOF), depth of anaesthesia monitoring (BIS) Anaesthesia induction: 1 mcg/kg fentanyl, 1 mg/kg lidocaine, 2-2.5 mg/kg propofol, 1 mg/kg rocuronium Intubation: It will be performed when BIS: 40-60, TOF rate is 0%. Right/left lateral position will be given according to the side of the patient's operation.

Before and after the surgical incision, the pre-emptive and postoperative block (ESPB / Paravertebral block) will be recorded from the side where the patient will be operated, at the T5 level, accompanied by routine USG.

Drug content to be administered*: total 25 cc volume (13.5 ml 0.5% bupivacaine + 5 ml 2% lidocaine + 1.5 ml morphine (morphine reconstituted with 0.9% NaCl to 1mg/ml) + 5 ml 0.9% NaCl) (This dose application is the routine doses applied in such surgeries in our clinic) Maintenance of anaesthesia: Desflurane : MAC titration with BIS in the range 40-60

Within the multimodal analgesia protocol:

1 mg/kg/h lidocaine infusion Dexketoprofen 50 mg iv 40 mg/kg Magnesium infusion (15 min in 100 cc 0.9% NaCl) Paracetamol 1 gram iv infusion (at the end of surgery) Anaesthetic drugs will be discontinued. 4mg/kg sugammadex will be administered to reverse neuromuscular blockade.

Extubation will be performed after BIS >90% and TOF ratio >90%. Postoperative intravenous PCA (patient controlled analgesia) will be prepared. PCA content: infusion: none -- bolus: 0.25 mcg/kg/min fentanyl -- lock time: 15 min Acute and chronic pain of the patients will be monitored in the postoperative period. (It will be evaluated with VAS (Visual analogue scale - ANNEX-1)).

Pain monitoring will be performed in the postoperative waking unit (20.min) and postoperative 2nd - 6th - 12th - 24th - 48th - 72nd hours.

The degree of pain at rest, with cough and movement (to be evaluated with VAS), the need for additional analgesics, the number of PCA bolus trials and the number given will be recorded. Postoperative oxygen requirement will be recorded.

Postoperative analgesia: IV Fentanyl PCA (Bolus 0.25 mcg/kg, locked time 15 minutes) If VAS >4 and PCA bolus is insufficient, parol 1 g iv or dexketoprofen 50 mg iv infusion is given.

For the evaluation of chronic pain, a phone call will be made at the 3rd month and 6th month postoperatively and pain questioning will be performed.

* Presence/absence of pain, VAS score if present, whether there is a need for chronic analgesics, whether there is a need for additional intervention, what was done if additional analgesic intervention was performed * Local anaesthetic drug doses in regional anaesthesia : source: Kirk, P. H. I. I. L. I. I. P. P., & Berde, C. B. (2020). Local anaesthetics. Miller's Anaesthesia. 9th ed. Philadelphia: Elsevier Inc, 878-9.

RANDOMİSATİON: The randomisation of the volunteers participating in the study will be ensured by randomising the order in which the patients were historically admitted to the operation and the method to be applied during the writing of the protocol.

After the study started, the groups were determined as follows by accepting the order in which the patients were historically admitted to the operation.

GROUP E: ESP group: 1,3,4,6,8,10, 14, 15, 17, 18, 22, 23, 24, 27, 28, 29, 32, 33, 36, 38, 44,45,46,47, 53, 54, 55, 56, 57, 58, 61, 64, 65, 68, 70, 72, 73, 76, 77

GROUP P: Paravertebral Group: 2, 5, 7, 9, 11,12, 13, 16, 19, 20, 21, 25,26,30,31, 34, 35, 37, 39, 40, 41, 42, 43, 48, 49, 50, 51, 52, 59, 60, 62, 63, 66, 67, 69, 71, 74, 75, 78

STATISTICAL ANALYSIS

* SAMPLE DIAMETER The sample size of the study was calculated in G*Power 3.1.9.2 programme. In the sample article, the mean PCA demand dose was 36.64±26.9 in the ESPB group and 18.82±13.67 in the TPVB group. When these data were taken into consideration, the effect size was calculated as 0.83, α=0.05 and 95% power and the sample size required for each group was calculated as 39 (total 78).
* STATISTICAL ANALYSIS Data will be analysed in IBM SPSS Statistics (version 23) package programme. Descriptive statistics will be shown as mean ± standard deviation for variables with normal distribution, median (min - max) for variables with non-normal distribution, number of cases and (%) for nominal variables.

The significance of the difference between the groups in terms of means will be investigated by t test and the significance of the difference in terms of median values will be investigated by mann whitney test. Nominal variables will be evaluated by Pearson Chi-Square or Fisher exact test.

In continuous variables, the change according to time before and after treatment will be investigated by paired t test if the distribution is normal and by Wilcoxon test if the distribution is not normal. When there are more than two follow-up times, the change will be investigated by repeated measures analysis of variance if the distribution is normal and Friedman test if the distribution is not normal. The change according to time, group and group*time interaction will be investigated by two-way analysis of variance in repeated measures if the distribution is normal, and by F1_LD_F1 nonparametric method if the distribution is not normal.

The results will be considered statistically significant for p<0.05.

At the end of the study, all eligible volunteers who completed the study will be included in the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* ASA I-II
* Patients with a VATS (video-assisted thoracic surgery) plan

Exclusion Criteria:

* Under 18 years old
* Patients under 40kg and BMI over 35
* Allergic to the drugs to be used in the study
* Patients with a history of chronic painkiller use
* Patients who refused to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Acute postoperative pain | 4 month
  Lower pain scores with erector spina plan block in pain control after acute thoracoscopy (using visual analogue scale, lowest value (no pain): 0, highest value (most severe pain): 10, lower values are considered as good results)

SECONDARY OUTCOMES:
Chronic postoperative pain | 6 month
  Less chronic pain with erector spinae block (using visual analogue scale, lowest value (no pain): 0, highest value (most severe pain): 10, lower values are considered as good results)

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University, Ankara, Altındağ, Turkey (Türkiye)

REFERENCES:
- [Background] Clairoux, A., Issa, R., Bélanger, M. È., Urbanowicz, R., Richebé, P., & Brulotte, V. (2023). Perioperative pain management for thoracic surgery: a narrative review of the literature. Current Challenges in Thoracic Surgery, 5.
- [Background] Makkad B, Heinke TL, Sheriffdeen R, Khatib D, Brodt JL, Meng ML, Grant MC, Kachulis B, Popescu WM, Wu CL, Bollen BA. Practice Advisory for Preoperative and Intraoperative Pain Management of Thoracic Surgical Patients: Part 1. Anesth Analg. 2023 Jul 1;137(1):2-25. doi: 10.1213/ANE.0000000000006441. Epub 2023 Apr 20. PMID 37079466
- [Background] Lin J, Liao Y, Gong C, Yu L, Gao F, Yu J, Chen J, Chen X, Zheng T, Zheng X. Regional Analgesia in Video-Assisted Thoracic Surgery: A Bayesian Network Meta-Analysis. Front Med (Lausanne). 2022 Apr 6;9:842332. doi: 10.3389/fmed.2022.842332. eCollection 2022. PMID 35463038
- [Background] Feray S, Lubach J, Joshi GP, Bonnet F, Van de Velde M; PROSPECT Working Group *of the European Society of Regional Anaesthesia and Pain Therapy. PROSPECT guidelines for video-assisted thoracoscopic surgery: a systematic review and procedure-specific postoperative pain management recommendations. Anaesthesia. 2022 Mar;77(3):311-325. doi: 10.1111/anae.15609. Epub 2021 Nov 5. PMID 34739134
- [Background] Batchelor TJP, Rasburn NJ, Abdelnour-Berchtold E, Brunelli A, Cerfolio RJ, Gonzalez M, Ljungqvist O, Petersen RH, Popescu WM, Slinger PD, Naidu B. Guidelines for enhanced recovery after lung surgery: recommendations of the Enhanced Recovery After Surgery (ERAS(R)) Society and the European Society of Thoracic Surgeons (ESTS). Eur J Cardiothorac Surg. 2019 Jan 1;55(1):91-115. doi: 10.1093/ejcts/ezy301. PMID 30304509
- [Background] Hamilton C, Alfille P, Mountjoy J, Bao X. Regional anesthesia and acute perioperative pain management in thoracic surgery: a narrative review. J Thorac Dis. 2022 Jun;14(6):2276-2296. doi: 10.21037/jtd-21-1740. PMID 35813725
- [Background] Shim JG, Ryu KH, Kim PO, Cho EA, Ahn JH, Yeon JE, Lee SH, Kang DY. Evaluation of ultrasound-guided erector spinae plane block for postoperative management of video-assisted thoracoscopic surgery: a prospective, randomized, controlled clinical trial. J Thorac Dis. 2020 Aug;12(8):4174-4182. doi: 10.21037/jtd-20-689. PMID 32944329
- [Background] Taketa Y, Irisawa Y, Fujitani T. Comparison of ultrasound-guided erector spinae plane block and thoracic paravertebral block for postoperative analgesia after video-assisted thoracic surgery: a randomized controlled non-inferiority clinical trial. Reg Anesth Pain Med. 2019 Nov 8:rapm-2019-100827. doi: 10.1136/rapm-2019-100827. Online ahead of print. PMID 31704789
- [Background] Zhao H, Xin L, Feng Y. The effect of preoperative erector spinae plane vs. paravertebral blocks on patient-controlled oxycodone consumption after video-assisted thoracic surgery: A prospective randomized, blinded, non-inferiority study. J Clin Anesth. 2020 Jun;62:109737. doi: 10.1016/j.jclinane.2020.109737. Epub 2020 Feb 21. PMID 32092617
- [Background] Chen N, Qiao Q, Chen R, Xu Q, Zhang Y, Tian Y. The effect of ultrasound-guided intercostal nerve block, single-injection erector spinae plane block and multiple-injection paravertebral block on postoperative analgesia in thoracoscopic surgery: A randomized, double-blinded, clinical trial. J Clin Anesth. 2020 Feb;59:106-111. doi: 10.1016/j.jclinane.2019.07.002. Epub 2019 Jul 19. PMID 31330457
- [Background] Turhan O, Sivrikoz N, Sungur Z, Duman S, Ozkan B, Senturk M. Thoracic Paravertebral Block Achieves Better Pain Control Than Erector Spinae Plane Block and Intercostal Nerve Block in Thoracoscopic Surgery: A Randomized Study. J Cardiothorac Vasc Anesth. 2021 Oct;35(10):2920-2927. doi: 10.1053/j.jvca.2020.11.034. Epub 2020 Nov 20. PMID 33358107
- [Background] Crile, G. (1913). The kinetic theory of shock and its prevention through anoci-association (shocklessoperation). The Lancet, 182(4688), 7-16.
- [Background] Woolf CJ. Evidence for a central component of post-injury pain hypersensitivity. Nature. 1983 Dec 15-21;306(5944):686-8. doi: 10.1038/306686a0. PMID 6656869
- [Background] Fuller AM, Bharde S, Sikandar S. The mechanisms and management of persistent postsurgical pain. Front Pain Res (Lausanne). 2023 Jul 6;4:1154597. doi: 10.3389/fpain.2023.1154597. eCollection 2023. PMID 37484030